CLINICAL TRIAL: NCT07378033
Title: A Randomized, Double-Blind, Placebo-Controlled Trial Evaluating the Safety and Efficacy of Cornfit™ for Body Fat Reduction and Weight Management
Brief Title: Body Fat Reduction and Weight Management
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Bioagile Therapeutics Pvt. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: BSP-25-075; CTRI/2025/10/095913 (Other: Clinical Trial Registry India)
Record Dates: First submitted 2026-01-02; First posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Obesity & Overweight
Keywords: Weight management
MeSH Terms: conditions — Obesity; Overweight | interventions — Dietary Supplements

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cornfit™ (Experimental): Corn silk (Stigma maydis)
  Interventions: Dietary Supplement: Dietary Supplement
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo Control

INTERVENTIONS:
Dietary Supplement: Dietary Supplement — active drug
  Arms: Cornfit™
Other: Placebo Control — placebo
  Arms: Placebo

SUMMARY:
Obesity is a chronic complex disease defined by excessive fat deposits that can impair health. Obesity can lead to increased risk of type 2 diabetes and heart disease, it can affect bone health and reproduction, it increases the risk of certain cancers. Obesity influences the quality of living, such as sleeping or moving. The diagnosis of overweight and obesity is made by measuring people's weight and height and by calculating the body mass index (BMI): weight kg/height² m². The body mass index is a surrogate marker of fatness and additional measurements, such as the waist circumference, can help the diagnosis of obesity. The BMI categories for defining obesity vary by age and gender in infants, children and adolescents. Corn silk also known as Stigma maydis is a type of agricultural waste composed of a long, silky, hair-like structure ranging from yellowish to reddish in colour. In vitro and in vivo studies of corn silk showed adipogenesis, lipid metabolism and body weight management. Additionally, it reduces and inhibits adipose tissue formation and reduces the size of adipocytes and prevents excess fat accumulation. The anti-obesity effect of maize silk extract decreases the absorption of dietary fat and suppresses the formation of fatty acids. Corn silk inhibits the expression of adipogenic transcription factors like the peroxisome proliferator-activated receptor gamma and CCAAT/enhancer-binding proteins C/EBPs and prevents the differentiation of pre-mature adipocytes into mature adipocytes, it also suppresses the development of adipose tissue and the accumulation of excess fat.

ELIGIBILITY:
Inclusion Criteria:

1. Adult males and non-pregnant females aged 19 to 65 years
2. Individuals with a BMI of 25-32kg/m2 who are not taking any obesity related medicines.
3. Able to comply with all required study procedures and schedule.
4. Able to comply and willing to follow the prescribed diet plan.
5. Willing and able to give written informed consent.

Exclusion Criteria:

1. Individuals who experienced a weight change of 5% or more within 3 months prior to the screening.
2. Individuals who have taken or used medications, herbal remedies, or health supplements (including probiotics) for anti- obesity purposes (e.g., energy metabolism, appetite suppression, weight control, fat breakdown, carbohydrate blocking, inhibition of fat absorption, or gastrointestinal activity regulation) within 6 months prior to the screening.
3. Individuals who have participated in or experienced a weight-loss program within 3 months prior to the screening.
4. Individuals with Gastrointestinal disease like Crohn's Disease, Inflammatory Bowel Syndrome, Gastric resection, Chronic Inflammation (Kidney, Liver, Pancreas), infectious diseases, Autoimmune diseases, Malabsorption syndrome, Porphyria, Hepatitis B or C carriers.
5. Individuals currently using immunosuppressants; proton pump inhibitors (PPIs), H2 receptor blockers, or nonsteroidal anti-inflammatory drugs (NSAIDs); insulin; thyroid hormone replacement therapy.
6. Individuals who have taken Appetite suppressants, Semaglutide, OTC weight loss supplements 3 to 6 months before the trial.
7. Individuals who have consistently consumed dietary supplements (including protein supplements), teas, beverages, or jellies for weight control or fat reduction purposes.
8. Individuals who have undergone any obesity surgery or any surgery within the last 6 months.
9. Individuals who have consistently taken medications or health supplements for cholesterol improvement or blood circulation enhancement within 6 months prior to the screening.
10. Individuals who have clinically significant diseases or disorders related to the liver, kidneys, pancreas, biliary system, cardiovascular system, respiratory system, endocrine system (e.g., diabetes, thyroid disorders), or central nervous system, or who have malignant tumors as identified in physical or clinical examinations (except those who have not experienced recurrence for over 5 years post-surgery).
11. Individuals with uncontrolled hypertension (systolic blood pressure greater or equal to 160 mmHg or diastolic blood pressure greater or equal to 100 mmHg).
12. Individuals diagnosed with diabetes and taking medications to control blood sugar.
13. Individuals undergoing psychiatric medication or psychotherapy for eating disorders or other mental disorders.
14. Individuals with a history of clinically significant hypersensitivity reactions or those who may exhibit hypersensitivity to the ingredients or similar components of the investigational product.
15. Individuals who have consistently used functional products for cellulite removal or fat breakdown.
16. Heavy smokers (greater or equal to 20 cigarettes/day).
17. Individuals who excessively consume alcohol (greater or equal to 40 g/day for men or greater or equal to20 g/day for women).
18. Individuals whose diagnostic or medical test results at the screening visit show the following AST, ALT, or gamma GTP levels exceeding three times the upper limit of the laboratory reference range. eGFR less 60 mL/min/1.73 m square.
19. Individuals who have participated in other clinical trials or human application studies within 3 months prior to the screening.
20. Pregnant or lactating women or within 6 months of giving birth
21. Individuals deemed unsuitable for participation in the study by the principal investigator based on diagnostic laboratory results or other reasons

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-10-23 (Actual); Primary Completion 2026-04-10 (Estimated); Study Completion 2026-05-10 (Estimated)

PRIMARY OUTCOMES:
Change in total body fat mass assessed by DEXA at 12 weeks | Day 0, Day 1, Day 42, Day 84
  Change in total body fat mass from baseline to Week 12, measured using dual-energy X-ray absorptiometry (DEXA), comparing the intervention and placebo groups

SECONDARY OUTCOMES:
Change in regional body fat mass by body area assessed by DEXA at 12 weeks | Day 0, Day 1, Day 42, Day 84
  Change in regional body fat mass from baseline to Week 12 in the whole body, arms, legs, trunk, android, and gynoid regions, measured using dual-energy X-ray absorptiometry (DEXA), comparing the intervention and placebo groups.
Change in total body fat percentage assessed by DEXA at 12 weeks | Day 0, Day 1, Day 42, Day 84
  Change in total body fat percentage from baseline to Week 12, measured using dual-energy X-ray absorptiometry (DEXA), comparing the intervention and placebo groups
Change in lean mass percentage assessed by DEXA at 12 weeks | Day 0, Day 1, Day 42, Day 84
  Change in lean mass percentage from baseline to Week 12, measured using dual-energy X-ray absorptiometry (DEXA), comparing the intervention and placebo groups.
Change in total abdominal fat area assessed by abdominal CT at 12 weeks | Day 0, Day 1, Day 42, Day 84
  Change in total abdominal fat area from baseline to Week 12, measured using abdominal computed tomography (CT), comparing the intervention and placebo groups.
Change in subcutaneous fat area assessed by abdominal CT at 12 weeks | Day 0, Day 1, Day 42, Day 84
  Change in subcutaneous fat area from baseline to Week 12, measured using abdominal computed tomography (CT), comparing the intervention and placebo groups.
Change in visceral fat area assessed by abdominal CT at 12 weeks | Day 0, Day 0, Day 42, Day 84
  Change in visceral fat area from baseline to Week 12, measured using abdominal computed tomography (CT), comparing the intervention and placebo groups.

CONTACTS AND LOCATIONS:
Overall Officials: Dr H N Shivaprasad Prasad, Study Director — Botanic Healthcare Private Limited
Locations (1):
- Raksha health care, Bangalore, Karnataka, India

IPD SHARING:
Plan to Share IPD: No